CLINICAL TRIAL: NCT01469299
Title: Prospective Study Measuring Clinical Outcomes of Knee Arthroplasty Using the VERASENSE™ Knee System
Status: Completed | Type: Observational
Sponsor: Orthosensor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1-Anderson
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthritis, Avascular Necrosis, Rheumatoid Arthritis, Post-traumatic Arthritis
Keywords: Ligament Balance, Total Knee Arthroplasty, Intra-operative Sensors
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objectives of this evaluation are: 1) To attempt to refine the current clinical understanding of "balance" 2) To determine if patients with quantifiably balanced knee joints exhibit improved clinical outcomes versus patient with residual imbalance, as measured by the VERASENSE™ Knee System

Secondary objectives:

* Determine whether a difference in inter-compartment loads and soft tissue tension exists between the physicians intra-operative feel compared to the quantifiable data measured by the VERASENSE™ Knee System
* Determine which ligament releases are performed by the surgeon to improve soft tissue balance while utilizing the information from the VERASENSE™ Knee System
* Evaluate range of motion, pain, physical function, activity level, and patient satisfaction between baseline (pre-operative) and post-operative follow-up as well as radiographic success and survivorship of the knee implants

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a candidate for a primary total knee replacement
* Subject must be diagnosed with one or more of the following conditions: osteoarthritis, avascular necrosis, rheumatoid or other inflammatory arthritis post-traumatic arthritis
* Subject's joint must be anatomically and functionally suited to receive the selected implant
* Subject is 50 years of age or older (≥ 50 yrs) at the time of consent
* Subject is likely to be available for all study visits
* Subject is able and willing to sign the informed consent and follow study procedures
* Subject is not pregnant

Exclusion Criteria:

* Prior total knee arthroplasty
* Subject has a mental condition that may interfere with the subject's ability to give an informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the Subject cannot understand the informed consent process, global dementia, prior strokes that interfere with the Subject's cognitive abilities, senile dementia, and Alzheimer's Disease)
* Subject is pregnant
* Subject has an active infection or joint sepsis
* Subject has muscular, neurological or vascular deficiencies which compromise the affected extremity (i.e., Parkinson's Disease, Multiple Sclerosis, and Charcot joints)
* Ligament insufficiencies, prior surgeries such as ACL or PCL reconstructions, posterolateral reconstructions, osteotomies, tibia plateau fractures
* Range of Motion less than 90 degrees, flexion contracture of more than 20 degrees

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2011-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Joint Balance | At time of Total Knee Surgery

SECONDARY OUTCOMES:
Patient Reported Outcome Measures | Changes from Baseline at 3-years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Gustke, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (8):
- United States (8):
  - St. Helena Hospital, St. Helena, California
  - Holy Cross Orthopedic Institute, Fort Lauderdale, Florida
  - Naples Community Hospital, Naples, Florida
  - Tampa General/FORE, Tampa, Florida
  - Emory Healthcare - St. Joseph's Research Institute, Atlanta, Georgia
  - Spectrum Health/Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Trinity Health/Bone and Joint Institute, Port Huron, Michigan
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- Available data/document: Publication — https://www.ncbi.nlm.nih.gov/pubmed/24269069 — 6-Month Report: Guske et al. A New Method for Defining Balance: Promising Short-term outcomes of Sensor-Guided TKA. J Arthroplasty. 2014 May;29(5):955-60
- Available data/document: Publication — https://www.ncbi.nlm.nih.gov/pubmed/25210632 — 1-year Report: Gustke et al. Primary TKA patients with Quantifiably Balanced Soft-Tissue Achieve Significant Clinical Gains Sooner than Unbalanced Patients. Adv Orthop. 2014:628695